CLINICAL TRIAL: NCT03019627
Title: An 8-week, Phase II, Single-center, Randomized, Double-masked, Vehicle-controlled, Parallel-group Study With 4 Weeks of Follow-up to Evaluate Safety and Efficacy of rhNGF Eye Drops Solution vs Vehicle in Patients With Dry Eye
Brief Title: An 8-week Study to Evaluate Safety and Efficacy of NGF Eye Drops Solution Versus Vehicle in Patients With Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NGF0216
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Nerve Growth Factor; cenegermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The identity of the treatments was concealed from the patient, Investigator, site staff, and Dompé's clinical research personnel until the study was unmasked for the final statistical analysis (after data base lock) except in case of specific events that required unmasking of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rhNGF 20μg/mL (Experimental): Recombinant Human Nerve Growth Factor (rhNGF) at 20 μg/mL eye drops six times daily
  Interventions: Drug: NGF
- Vehicle (Placebo Comparator): vehicle eye drops six times daily
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: NGF — Eye Drop 20 μg/mL
  Other Names: cenegermin
  Arms: rhNGF 20μg/mL
Other: Vehicle — Vehicle Eye Drop
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
The primary objective of this study was to assess the efficacy and safety of rhNGF when administered as eye drops to patients with dry eye

The secondary objectives of this study were:

* To assess change from baseline in Symptom Assessment In Dry Eye (SANDE) scores (without imputation), corneal and conjunctival staining according to National Eye Institute (NEI) scale, and in Tear Film Break-up Time (TFBUT) and Schirmer test I, following 4 and 8 weeks of treatment.
* To assess change in levels of inflammatory biomarker matrix metallopeptidase 9 (MMP-9) in tears following 8 weeks of treatment.
* To assess the incidence and frequency of treatment-emergent adverse events (TEAEs) following 8 weeks of treatment.

DETAILED DESCRIPTION:
The proposed phase II study is a single-center, randomized, double-masked, parallel-arm, vehicle-controlled trial, designed to evaluate the safety and efficacy of Recombinant Human Nerve Growth Factor (rhNGF) eye drops at 20 μg/ml concentration administered six times daily for 8 weeks in patients with dry eye. After confirmation of inclusion and exclusion criteria all eligible patients will be randomized at 2:1 ratio to rhNGF or vehicle control treatment with 8 weeks of study treatments administration with 4 weeks Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male or female) must be ≥ 18 years of age.
2. Patients must be diagnosed with any type of dry eye (e.g. Meibomian Gland Dysfunction, Blepharitis, Keratoconjunctivitis sicca etc) at least 3 months before enrollment.
3. Patients must present dry eye pathology characterized by the following clinical features:

   1. Corneal and/or conjunctival staining with fluorescein and lissamine green using National Eye Institute (NEI) grading system > 3
   2. Mean Symptom Assessment in Dry Eye (SANDE) questionnaire ≥30
   3. Schirmer test without anesthesia < 10 mm/5 minutes and/or tear film break-up time (TFBUT) < 10 seconds in the study eye
4. The same eye (study eye) must fulfill all the above criteria.
5. Patients must have best corrected distance visual acuity (BCDVA) score of ≥ 0.1 decimal units in both eyes at the time of study enrollment.
6. Female patients must have negative pregnancy test if at childbirth potential.
7. Only patients who satisfy all requirements for informed consent may be included in the study. Written Informed Consent must be obtained before the initiation of any study specific procedures.
8. Patients must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

1. Best corrected distance visual acuity (BCDVA) score of < 0.1 decimal units in either eye.
2. Evidence of an active ocular infection in either eye.
3. Presence or history of any ocular disorder or condition, including ocular surgery, trauma, or disease that could possibly interfere with the interpretation of study results in the opinion of the Investigator.
4. Intraocular inflammation defined as Tyndall score >0.
5. Active or recent diagnosis of malignancy (i.e., currently under chemo/radiotherapy).
6. Systemic disease not stabilized within 1 month before baseline visit (e.g., uncontrolled diabetes; thyroid malfunction) or judged by the Investigator to be incompatible with the study (e.g., current systemic infections) or with a condition incompatible with the frequent assessment required by the study.
7. Patients who have had a serious adverse reaction or significant hypersensitivity to any drug or chemically related compounds, or had a clinically significant allergy to drugs, foods, amide local anesthetics, or other materials, including commercial artificial tears containing carboxymethylcellulose (CMC) (in the opinion of the Investigator).
8. Use of topical cyclosporine, topical corticosteroids, or any other topical medication for the treatment of dry eye in either eye until the day of study enrollment.
9. Contact lenses or punctal plug use during the study (previous use not an exclusion criteria, but must be discontinued at the baseline visit.
10. An anticipated need of additional systemic treatments for dry eye during the study (all prior treatment must be continued for the entire duration of the study).
11. Females of childbearing potential (those who are not surgically sterilized or postmenopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

    1. are currently pregnant or,
    2. have a positive result at the urine pregnancy test (Baseline/Day 0) or,
    3. intend to become pregnant during the study treatment period or,
    4. are breast-feeding or,
    5. are not willing to use highly effective birth control measures, such as: hormonal contraceptives - oral, implanted, transdermal, or injected - and/or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or a intrauterine device (IUD) - during the entire course of and 30 days after the study treatment periods.
12. History of drug addiction or alcohol abuse.
13. Any prior ocular surgery (including refractive palpebral and cataract surgery) if within 90 days before the screening visit.
14. Participation in a clinical trial with a new active substance during the past 30 days.
15. Participation in another clinical trial study at the same time as the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomina Massaro Giordano, MD, Principal Investigator — Penn Dry Eye and Oc. Surf. Center, Univ. of Pennsylvania, Scheie Eye Institute
Locations (1):
- Penn Dry Eye and Ocular Surface Center, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After confirmation of inclusion and exclusion criteria all eligible patients were randomized at 2:1 ratio to rhNGF or vehicle control treatment with 8 weeks of study treatments administration with 4 weeks Follow-up. rhNGF and vehicle were administered as eye drops at 20 μg/mL concentration, six times daily for 8 weeks in patients with dry eye
Period: Overall Study
Arm/Group | rhNGF 20μg/mL | Vehicle
Started | 100 | 50
Completed | 85 | 42
Not Completed | 15 | 8
Not completed — Adverse Event | 8 | 0
Not completed — Unrelated to adverse event | 1 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — not compliance | 2 | 2
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Enrolled set = All patients who were randomized comprised the Enrolled Set. Data from this set was used to summarize demographic, baseline, and background characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | rhNGF 20μg/mL | Vehicle | Total
Number analyzed (Participants) | 100 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (11.89) | 57.7 (10.33) | 57.5 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 46 | 131
  Male | 15 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 99 | 48 | 147
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 50 | 150
Number of baseline participants [Count of Participants; unit: Participants] | 100 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Symptom Assessment in Dry Eye (SANDE) Scores
Description: Change from baseline with Last Observation Carried Forward (LOCF) imputation. LOCF is a method of imputing missing data in longitudinal studies and tests for difference in mean rates of change in controlled repeated measurements designs with dropouts.
  The SANDE score is calculated by taking the square root of the product of the frequency of symptoms score and the severity of symptoms score. The SANDE scale ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms.
Time Frame: week 8
Population: Full analysis set population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rhNGF 20μg/mL | Vehicle
Number analyzed (Participants) | 97 | 48
units on a scale
  Frequency: number analyzed (Participants) | 96 | 48
  Frequency | -38.8 (28.97) | -34.0 (26.67)
  Severity | -32.2 (31.04) | -31.07 (28.32)
Statistical Analysis 1: Comparison: rhNGF 20μg/mL vs Vehicle; Frequency statistical analysis; Test type: Superiority; p = 0.428, ANCOVA; difference in least square means = -3.83, 95% CI 2-sided [-13.34 to 5.68]
Statistical Analysis 2: Comparison: rhNGF 20μg/mL vs Vehicle; Severity statistical analysis; Test type: Superiority; p = 0.974, ANCOVA; difference in least square means = 0.16, 95% CI 2-sided [-9.45 to 9.76]

2. Secondary Outcome: SANDE Scores
Description: as for outcome 1
Time Frame: Week 4, week 8, week 12
Population: Full analysis set population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rhNGF 20μg/mL | Vehicle
Number analyzed (Participants) | 97 | 48
units on a scale
  Frequency - week 4: number analyzed (Participants) | 94 | 47
  Frequency - week 4 | -22.1 (24.08) | -20.4 (20.66)
  Frequency - week 8: number analyzed (Participants) | 86 | 42
  Frequency - week 8 | -39.6 (28.55) | -34.6 (27.60)
  Frequency - week 12: number analyzed (Participants) | 88 | 42
  Frequency - week 12 | -44.8 (28.69) | -28.2 (28.94)
  Severity - week 4: number analyzed (Participants) | 94 | 47
  Severity - week 4 | -19.9 (25.20) | -22.2 (24.31)
  Severity - week 8: number analyzed (Participants) | 86 | 42
  Severity - week 8 | -32.6 (30.64) | -33.1 (28.30)
  Severity - week 12: number analyzed (Participants) | 88 | 42
  Severity - week 12 | -38.8 (29.20) | -24.3 (28.43)
Statistical Analysis 1: Comparison: rhNGF 20μg/mL vs Vehicle; frequency statistical analysis - week 4; Test type: Superiority; p = 0.783, ANCOVA; Difference in least square means = -1.12, 95% CI 2-sided [-9.14 to 6.91]
Statistical Analysis 2: Comparison: rhNGF 20μg/mL vs Vehicle; Frequency statistical analysis - week 8; Test type: Superiority; p = 0.461, ANCOVA; difference in least square means = -3.82, 95% CI 2-sided [-14.1 to 6.41]
Statistical Analysis 3: Comparison: rhNGF 20μg/mL vs Vehicle; Frequency statistical analysis - week 12; Test type: Superiority; p = 0.004, ANCOVA; difference in least square means = -15.3, 95% CI 2-sided [-25.6 to -4.97]
Statistical Analysis 4: Comparison: rhNGF 20μg/mL vs Vehicle; Severity statistical analysis - week 4; Test type: Superiority; p = 0.544, ANCOVA; difference in least square means = 2.55, 95% CI 2-sided [-5.72 to 10.82]
Statistical Analysis 5: Comparison: rhNGF 20μg/mL vs Vehicle; Severity statistical analysis - week 8; Test type: Superiority; p = 0.837, ANCOVA; difference in least square means = 1.06, 95% CI 2-sided [-9.12 to 11.24]
Statistical Analysis 6: Comparison: rhNGF 20μg/mL vs Vehicle; Severity statistical analysis - week 12; Test type: Superiority; p = 0.007, ANCOVA; difference in least square means = -13.8, 95% CI 2-sided [-23.7 to 3.88]

3. Secondary Outcome: Cornea Vital Staining
Description: Changes from baseline on National Eye Institute (NEI) scale. The NEI/Industry Workshop guidelines were used for grading the scale of corneal and conjunctival damage. The cornea was divided into five sectors (central, superior, inferior, nasal and temporal), each of which was scored on a scale of 0-3, with a maximal total corneal staining score of 15.
  Both nasally and temporally, the conjunctiva was divided into a superior paralimbal area, an inferior paralimbal area, and a peripheral area with a grading scale of 0-3 and with a maximal total score of 9 for the nasal and temporal conjunctiva (overall the total score ranged from 0-18).
  Briefly, grade 0 reflected normal/healthy situation, whereas grade 3 reflected a severe damage in the considered sector.
Time Frame: week 4, week 8, week 12
Population: Full analysis set population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rhNGF 20μg/mL | Vehicle
Number analyzed (Participants) | 97 | 48
units on a scale
  week 4: number analyzed (Participants) | 94 | 47
  week 4 | -3.5 (2.32) | -3.0 (2.27)
  week 8: number analyzed (Participants) | 86 | 41
  week 8 | -4.2 (2.92) | -4.4 (2.70)
  week 12: number analyzed (Participants) | 88 | 42
  week 12 | -4.4 (2.80) | -5.1 (2.93)
Statistical Analysis 1: Comparison: rhNGF 20μg/mL vs Vehicle; week 4; Test type: Superiority; p = 0.046, ANCOVA; Difference in least square means = -0.70, 95% CI 2-sided [-1.38 to -0.01]
Statistical Analysis 2: Comparison: rhNGF 20μg/mL vs Vehicle; week 8; Test type: Superiority; p = 0.425, ANCOVA; Difference in least square means = -0.30, 95% CI 2-sided [-1.05 to 0.44]
Statistical Analysis 3: Comparison: rhNGF 20μg/mL vs Vehicle; week 12; Test type: Superiority; p = 0.788, ANCOVA; Difference in least square means = -0.09, 95% CI 2-sided [-0.76 to 0.58]

4. Secondary Outcome: Conjunctival Vital Staining
Description: as for outcome 3
Time Frame: week 4, week 8, week 12
Population: Full analysis set population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rhNGF 20μg/mL | Vehicle
Number analyzed (Participants) | 97 | 48
units on a scale
  week 4: number analyzed (Participants) | 94 | 47
  week 4 | -4.7 (3.94) | -4.1 (3.45)
  week 8: number analyzed (Participants) | 86 | 42
  week 8 | -6.7 (4.16) | -5.9 (4.07)
  week 12: number analyzed (Participants) | 88 | 42
  week 12 | -7.2 (4.23) | -7.0 (3.90)
Statistical Analysis 1: Comparison: rhNGF 20μg/mL vs Vehicle; week 4; Test type: Superiority; p = 0.265, ANCOVA; Difference in least square means = -0.71, 95% CI 2-sided [-1.95 to 0.54]
Statistical Analysis 2: Comparison: rhNGF 20μg/mL vs Vehicle; week 8; Test type: Superiority; p = 0.026, ANCOVA; Difference in least square means = -1.38, 95% CI 2-sided [-2.59 to -0.17]
Statistical Analysis 3: Comparison: rhNGF 20μg/mL vs Vehicle; week 12; Test type: Superiority; p = 0.361, ANCOVA; Difference in least square means = -0.60, 95% CI 2-sided [-1.90 to 0.70]

5. Secondary Outcome: Change in Tear Film Break-up Time (TFBUT)
Description: TFBUT was measured by determining the time to tear break-up. The TFBUT was performed after instillation of 5 μL of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. The patient was instructed to blink several times to thoroughly mix the fluorescein with the tear film.
Time Frame: week 4, week 8, week 12
Population: Full analysis set population
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | rhNGF 20μg/mL | Vehicle
Number analyzed (Participants) | 97 | 48
seconds
  week 4: number analyzed (Participants) | 94 | 47
  week 4 | 0.4 (1.68) | 0.8 (1.57)
  week 8: number analyzed (Participants) | 86 | 42
  week 8 | 0.5 (1.74) | 0.7 (1.89)
  week 12: number analyzed (Participants) | 88 | 42
  week 12 | 0.5 (2.34) | 0.9 (1.42)
Statistical Analysis 1: Comparison: rhNGF 20μg/mL vs Vehicle; week 4; Test type: Superiority; p = 0.323, ANCOVA; Difference in least square means = -0.25, 95% CI 2-sided [-0.76 to 0.25]
Statistical Analysis 2: Comparison: rhNGF 20μg/mL vs Vehicle; week 8; Test type: Superiority; p = 0.908, ANCOVA; Difference in least square means = 0.03, 95% CI 2-sided [-0.55 to 0.62]
Statistical Analysis 3: Comparison: rhNGF 20μg/mL vs Vehicle; week 12; Test type: Superiority; p = 0.702, ANCOVA; Difference in least square means = -0.12, 95% CI 2-sided [-0.76 to 0.52]

6. Secondary Outcome: Change From Baseline in Wetting Distance
Description: The Schirmer test without anesthesia was performed to measure aqueous tear secretion prior to the instillation of any dilating or eye drops
Time Frame: week 8
Population: Full analysis set population
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | rhNGF 20μg/mL | Vehicle
Number analyzed (Participants) | 85 | 42
millimeters | 2.4 (11.41) | -3.1 (8.66)
Statistical Analysis 1: Comparison: rhNGF 20μg/mL vs Vehicle; Test type: Superiority; p = 0.003, ANCOVA; Difference in least square means = 5.75, 95% CI 2-sided [2.02 to 9.48]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each time point of the study (ie. Baseline visit, Week 4, Week 8 and ETV or early termination
Arm/Group | rhNGF 20μg/mL | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/50
Serious Adverse Events (participants affected / at risk) | 5/100 | 0/50
Other Adverse Events (participants affected / at risk) | 97/100 | 38/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 20μg/mL (N=100) | Vehicle (N=50)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 20μg/mL (N=100) | Vehicle (N=50)
Ocular discomfort (Eye disorders) | 69 (87) | 10 (17)
Eye pain (Eye disorders) | 42 (67) | 4 (4)
Eye irritation (Eye disorders) | 15 (19) | 10 (11)
Vision blurred (Eye disorders) | 13 (14) | 4 (6)
Photophobia (Eye disorders) | 12 (14) | 3 (3)
Eye pruritus (Eye disorders) | 8 (8) | 5 (5)
Eye discharge (Eye disorders) | 9 (13) | 1 (2)
Eyelid disorder (Eye disorders) | 8 (8) | 0 (0)
Eyelid oedema (Eye disorders) | 4 (6) | 1 (3)
Dry eye (Eye disorders) | 4 (4) | 1 (1)
Eyelid pain (Eye disorders) | 5 (5) | 0 (0)
Lacrimation increased (Eye disorders) | 3 (3) | 2 (2)
Ocular hyperaemia (Eye disorders) | 3 (8) | 1 (1)
Blepharospasm (Eye disorders) | 2 (3) | 2 (2)
Eye swelling (Eye disorders) | 4 (5) | 0 (0)
Eyelid margin crusting (Eye disorders) | 2 (2) | 1 (2)
Foreign body sensation in eyes (Eye disorders) | 3 (4) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 2 (2)
Eyelid pruritus (Eye disorders) | 2 (4) | 0 (0)
Asthenopia (Eye disorders) | 2 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 1 (1)
Eye allergy (Eye disorders) | 2 (2) | 0 (0)
Scleral haemorrhage (Eye disorders) | 1 (1) | 1 (1)
visual impairment (Eye disorders) | 2 (2) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 1 (1)
Eye paraesthesia (Eye disorders) | 1 (3) | 0 (0)
Conjunctival deposit (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Corneal oedema (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Eyelid irritation (Eye disorders) | 1 (1) | 0 (0)
Eyelid sensory disorder (Eye disorders) | 1 (1) | 0 (0)
Lacrimation decreased (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Scleral discolouration (Eye disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 12 (14) | 5 (11)
Migrane (Nervous system disorders) | 3 (3) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Autonomic failure syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cervical Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy idiopathic progressive (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 8 (10) | 5 (5)
Sinusitis (Infections and infestations) | 2 (2) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Generalized oedema (General disorders) | 0 (0) | 1 (1)
Humidity intolerance (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 1 (1) | 0 (0)
abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye burns (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 0 (0)
Hypersensivity (Immune system disorders) | 1 (2) | 0 (0)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 1 (1) | 0 (0)
Dental implantation (Surgical and medical procedures) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Eye laser surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhoid operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Vena cava filter removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Vein disorder (Vascular disorders) | 1 (1) | 0 (0)
Intraocular pressure test (Investigations) | 1 (1) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
LImitations and caveats are not specified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03019627/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT03019627/SAP_001.pdf